CLINICAL TRIAL: NCT01303991
Title: A Phase I Feasibility Study of Hexvix Photodynamic Therapy in Patients With Intermediate or High-risk Bladder Cancer
Brief Title: Hexvix Photodynamic Therapy in Patients With Bladder Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Photocure (Industry)
Collaborators: Karl Storz (Unknown)
Responsible Party: Photocure ASA
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PC B251/03
Record Dates: First submitted 2011-02-18; First posted 2011-02-25 (Estimated); Last update posted 2011-02-25 (Estimated); Status verified 2011-02

CONDITIONS: Intermediate or High-risk Bladder Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hexvix PDT (Experimental)
  Interventions: Other: Hexvix PDT with Karl Storz T-Light

INTERVENTIONS:
Other: Hexvix PDT with Karl Storz T-Light

SUMMARY:
The purpose of the study is to investigate the safety and feasibility of Hexaminolevulinate based photodynamic therapy in patients with intermediate or high-risk transitional cell carcinoma of the bladder.

DETAILED DESCRIPTION:
Non-muscle invasive bladder cancer is currently treated by transurethral resection (TURB) and/or fulguration. However, recurrence and progression rates following endoscopic treatment of visible lesions are significant. To prevent recurrent and progressive disease, adjuvant intravesical chemotherapy and immunotherapy are applied. There is also increasing interest in new therapeutic strategies such as photodynamic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 years or above who have given written informed consent.
* Patients with intermediate or high-risk superficial bladder cancer, defined as low-grade early recurrence within 6 months after local chemotherapy or BCG, primary or recurrent high-grade disease (TaG3, TaG3 with CIS or CIS alone) or patients with primary T1G3 who are tumour free at second resection.

Exclusion Criteria:

* Patients with muscle invasive tumour
* Patients with bladder shrinkage
* Patients who have received prior PDT for bladder cancer
* History of T1G3 disease or other indications for cystectomy
* Patient with porphyria
* Gross haematuria. (Note: Gross haematuria is defined as a heavy bladder bleed resulting in marked amounts of blood in the urine, which may interfere with PDT)
* Patients who have received BCG or chemotherapy within three months prior to Hexvix instillation, except for a single dose of chemotherapy for prevention of seeding after resection
* Known allergy to hexaminolevulinate or a similar compound
* Participation in other clinical studies either concurrently or within the last 30 days
* Women of child-bearing potential.
* Conditions associated with a risk of poor protocol compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2005-03; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events
  To assess the safety of photodynamic therapy (PDT) using Hexvix and the Karl Storz T-light PDT System in patients with recurrent bladder cancer.
  (assessment of adverse events, blood biochemistry, vital signs, urodynamics)

SECONDARY OUTCOMES:
The number of tumour-free patients after 6 months
  To assess the efficacy of Hexvix PDT in patients with intermediate and high-risk bladder cancer

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Zaak, MD, Principal Investigator — Urology Department, Medizinische Fakultät der LMU Muenchen